CLINICAL TRIAL: NCT02297555
Title: ENDOBARRIER® vs Conventional Therapy in the Management of Metabolic Syndrome in Obese Patients. Medico-economic Analysis as Part of a Randomized Controlled Multicenter Trial - ENDOMETAB
Brief Title: ENDOBARRIER® and Conventional Therapy in the Management of Metabolic Syndrome in Obese Patients
Acronym: ENDOMETAB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013_26; 2013-A00980-45 (Other: ID-RCB number, ANSM); STIC 2012 (Other: STIC number, Ministry of Health France)
Record Dates: First submitted 2014-09-18; First posted 2014-11-21 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Metabolic Syndrome
Keywords: Obesity; Metabolic Syndrome; ENDOBARRIER®
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional medical therapy (No Intervention): Conventional medical therapy is defined as the use of the latest lifestyle guidelines to optimize weight loss and glycaemic management, frequent home monitoring/titration strategies, use of latest approved drug therapy for treatment of hyperglycaemia and restoration of pancreatic B cell function, also for dyslipidemia and hypertension in addition to regular follow-up visits to a medical doctor from a multidisciplinary team
- ENDOBARRIER® (Experimental): The interventional therapy will be the device ENDOBARRIER® over conventional medical therapy
  Interventions: Device: ENDOBARRIER®

INTERVENTIONS:
Device: ENDOBARRIER® — This medical device consists of a tube (impermeable fluoropolymer) inserted endoscopically and secured by hooks in the wall of the duodenal bulb. From the anchor site, this duodeno-jejunal sheath covers 60 cm in the small intestine. It thus limits the contact of nutrients with digestive juices (bile and pancreatic juice) and initial absorption, at least in part mimicking duodenal exclusion of the gastric bypass, one of the techniques of bariatric surgery.
  Arms: ENDOBARRIER®

SUMMARY:
Obesity and metabolic syndrome (MS) are closely interrelated leading to increased mortality, mainly due to cardiovascular disease. In addition, some cancers are much higher when obesity is associated with metabolic syndrome. Bariatric surgery allows significant and sustained weight loss with marked improvement of MS. Considered too invasive, surgery is proposed to a small proportion of patients who could theoretically benefit. The ENDOBARRIER® device implanted endoscopically is an innovative approach developed for management of obesity in the non-surgical manner with benefits for improvement in MS already reported in literature.

DETAILED DESCRIPTION:
Obesity, defined as a body mass index (BMI) over 30 kg / m², has now affected more than 14% of the French population. This condition is associated with several co-morbidities, and increased mortality, mainly due to cardiovascular disease and some cancers. These risks are much higher when obesity is associated with metabolic syndrome.

Conventional medical care for metabolic syndrome, even conducted by multidisciplinary teams combining dietary advice, physical activity and psychological treatment offers only limited results, both in weight reduction and comorbidities. Bariatric surgery allows however a significant and sustained weight loss in the majority of cases, and a decrease in the frequency and severity of co-morbidities, including type 2 diabetes, and decreased mortality including cardiovascular. Considered too invasive by many practitioners and patients, surgery is therefore proposed to a small proportion of patients who could theoretically benefit.

The results of surgery have, however, validated the principle of the interventional treatment of obesity and its metabolic complications.

Different techniques that may replace surgery are currently being developed. Among these new approaches, the most successful is the device "endoluminal liner ENDOBARRIER®" (GI Dynamics ™, Boston, USA). The ENDOBARRIER® device could represent a major innovation in the non-surgical management of obesity. The benefits of installing the device on the morbidity associated with obesity are reported in the literature: impact on hypertension, diabetes, dyslipidemia and metabolic syndrome as such.

This trial will compare in a randomized study the results, tolerance and cost of the interventional therapy with the device ENDOBARRIER® over conventional therapy in French patients with obesity and metabolic syndrome, with or without diabetes. The evaluation of the cost-effectiveness of this device will clarify its role in the strategy for the management of obesity and its comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Metabolic Syndrome defined by the presence of at least 3 of the 5 factors identified in the harmonization of the definition of metabolic syndrome by the International Diabetes Federation, the American Heart Association and the National Heart, Lung and Blood Institute
* BMI > 30 kg/m2
* The subject must be a candidate for general anesthesia
* The subject must be able to understand the options to comply with the requirement of each intervention program.
* Non-pregnant female patients must agree to use a reliable method of contraception for 2 years

Exclusion Criteria:

* Contraindications from the notice of ENDOBARRIER device

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-04; Primary Completion 2017-01 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Frequency of patients without Metabolic Syndrome | 12 month
  The primary end point will be the rate of resolution of Metabolic Syndrome at 1 year as measured by frequency of patients without MS at 12 months.

SECONDARY OUTCOMES:
The level of insulin resistance | 12 months, 24 months
Changed in cardiovascular risk assessed by Framingham Risk Score | 12 months, 24 months
Changed in quality of life | 12 months, 24 months
Rate of adverse events | 12 months, 24 months
The cost-benefit ratio for each group | 12 months, 24 months
  The cost-benefit ratio for each group by evaluating the medical costs in each arm
Changed in blood pressure | 12 months, 24 months
  Changed in specific metabolic syndrome parameters such blood pressure
Changed in blood sugar | 12 months, 24 months
  Changed in blood sugar
Changed in triglycerides | 12 months, 24 months
  Changed in triglycerides
Changed in HDL | 12 months, 24 months
  Changed in HDL
Changed in waist circumference | 12 months, 24 months
  Changed in waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: François PATTOU, Professor, Principal Investigator — University Hospital of Lille
Locations (10):
- France (10):
  - Hôpital Avicenne, Bobigny
  - Hopital Ambroise Pare (Ap-Hp), Boulogne-Billancourt
  - Hopital Louis Mourier, Colombes
  - University Hospital Lille, Lille
  - Hospice civils de Lyon, Lyon
  - Assistance Publique des Hôpitaux de Marseille, Marseille
  - Centre Hospitalier Universitaire, Montpellier
  - Centre Hospitalier Universitaire, Nantes
  - Nouvel Hôpital Civil, Strasbourg
  - Hopital Larrey- Chu, Toulouse